CLINICAL TRIAL: NCT05958927
Title: Fundus Findings and Thiol-Disulfide Homeostais in Gestational Diabetes
Brief Title: Fundus Findings and Thiol-Disulfide Homeostais
Status: Completed | Type: Observational
Sponsor: Suzan Dogruya (Other)
Responsible Party: Sponsor-Investigator, Suzan Dogruya, Doctor, Uşak University
Organization: Uşak University (Other)
Other Study IDs: Gestational Diabetes
Record Dates: First submitted 2023-07-03; First posted 2023-07-25 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes; Eye Diseases; Retinal Disease; Oxidative Stress
MeSH Terms: conditions — Diabetes, Gestational; Eye Diseases; Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Non diabetic women
  Interventions: Other: tear test and eye measurement
- Case group: Women with impairment glucose status
  Interventions: Other: tear test and eye measurement

INTERVENTIONS:
Other: tear test and eye measurement — tear test and eye measurement

SUMMARY:
Gestational diabetes mellitus is associated with abnormal blood sugar levels throughout pregnancy in women without prior diabetes. Many studies have been conducted on the relationship between diabetes and oxidative stress. In this study, it was aimed to investigate the presence of fundus findings in patients with gestational diabetes and/or impaired blood sugar based on the results of previous studies and to simultaneously investigate the thiol-disulfide homeostasis in the tears of the patients.There was no previous study in the literature on thiol disulfide homeostasis in tears in gestational diabetic patients.

DETAILED DESCRIPTION:
This is a prospective case-control study conducted in 26 pregnant patients diagnosed with gestational diabetes at 24-28 weeks of pregnancy and 34 healthy pregnant women without gestational diabetes in the Uşak Training and Research Hospital Gynecology and Ophthalmology clinic. Glucose tolerance test; If the plasma glucose was 140 mg/dl or higher in the 1st hour after an oral 50 g glucose load, 100 g glucose was added after 8 hours of fasting. The result of 100 gr OGTT was evaluated according to Carpenter and Coustan criteria. Gestational diabetes was diagnosed if two or more of the four glucose levels were abnormal according to the Carpenter and Coustan criteria. Gestational diabetes was diagnosed if the plasma glucose level was 200 mg and above in pregnant women who were loaded with 50 g glucose.

A total of 60 pregnant women participated in the study. (26 gestational diabetes and 34 healthy pregnant women). Investigators excluded patients with type 1diabetes mellitus and type 2 diabetes mellitus, patient that history of ocular surface disease, topical/systemic medical therapy,with ocular inflamatuar disease such as üveitis. The patients who is healthy pregnant and gestasional diabetes mellitus pregnant were recruit to this study. Controls group included only healthy pregnant.

Tears analysis is less invasive, safe and accaptable method for research

All patients underwent a comprehensive ophthalmologic examination that included best-corrected visual acuity, slit-lamp examination, dilated fundus examination and applanation tonometry. Based on the International Clinical DR Disease Severity Scale (ICDRS).

Tears analysis is less invasive, safe and accaptable method for research. Tear samples, Schirmer paper strips were placed in the lower conjunctival fornix of the right eye for a maximum of 5 minutes. Care was taken not to use tear stimulation, topical anesthetic or other eye drops. Attention was paid to factors such as lighting and room temperature. The ocular surface was not damaged. Tear samples were collected by a single individual (SD). A 15-20 mm test result was considered as enough for biochemical analysis. Schirmer strips were diluted with 500 μl previously cooled PBS (phosphate-buffered saline), and stored in Eppendorf tubes until analysis (-80 °C).

At the end of the study, fundus findings and tear oxidative stress values of both groups will be compared.ELISA method will be used for determination of tear oxidative stress findings.

The study followed the tenets of the declaration of Helsinki and was approved by the Uşak üniversitesi Ethics Committee (13.04.2023 / 93-93-04). Written and informed con-sent of participants was obtained for each patient prior to the study.

ELIGIBILITY:
Example:

Inclusion Criteria:

* Healthy pregnant at 24-28 weeks of pregnancy
* Pregnant patients diagnosed with gestational diabetes and/or impaired blood sugar at 24-28 weeks of pregnancy

Exclusion Criteria:

* Type 1diabetes mellitus,
* Type 2 diabetes mellitus,
* Patient that history of ocular surface disease,
* Topical/systemic medical therapy with ocular inflamatuar disease such as üveitis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 60 pregnant women participated in the study. (30 gestational diabetes and/or impaired blood sugar and 30 healthy pregnant women).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Doğruya, Principal Investigator — Usak University Medical Faculty
Locations (1):
- Usak University Medical Faculty, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rask-Madsen C, King GL. Kidney complications: factors that protect the diabetic vasculature. Nat Med. 2010 Jan;16(1):40-1. doi: 10.1038/nm0110-40. No abstract available. PMID 20057426
- [Background] Barbour LA. New concepts in insulin resistance of pregnancy and gestational diabetes: long-term implications for mother and offspring. J Obstet Gynaecol. 2003 Sep;23(5):545-9. doi: 10.1080/0144361031000156500. No abstract available. PMID 12963518
- [Background] Karacay O, Sepici-Dincel A, Karcaaltincaba D, Sahin D, Yalvac S, Akyol M, Kandemir O, Altan N. A quantitative evaluation of total antioxidant status and oxidative stress markers in preeclampsia and gestational diabetic patients in 24-36 weeks of gestation. Diabetes Res Clin Pract. 2010 Sep;89(3):231-8. doi: 10.1016/j.diabres.2010.04.015. PMID 20537747
- [Background] Lopez-Tinoco C, Roca M, Garcia-Valero A, Murri M, Tinahones FJ, Segundo C, Bartha JL, Aguilar-Diosdado M. Oxidative stress and antioxidant status in patients with late-onset gestational diabetes mellitus. Acta Diabetol. 2013 Apr;50(2):201-8. doi: 10.1007/s00592-011-0264-2. Epub 2011 Feb 17. PMID 21327985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Pre-assignment Details: women with impaired glucose status and normal glucose status
Period: Overall Study
Arm/Group | Control Group | Case Group
Started | 34 (This study started April 2023) | 26 (This study started April 2023)
Completed | 34 (This study completed February 2024) | 26 (This study completed February 2024)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: control and case group (women with impaired glucose status) will undergo tear test and eye measurements
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Case Group | Total
Number analyzed (Participants) | 34 | 26 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Women between the ages of 18 and 40 years
  years | 25.94 (4.50) | 28.30 (4.81) | 27.05 (4.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 26 | 60
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Turkish women were involved in this study
  Participants | 34 | 26 | 60
Region of Enrollment [Count of Participants; unit: Participants] — case control study, observational
  Participants
    Turkey | 34 | 26 | 60
oxidative stress markers [Mean (Standard Deviation); unit: mmol/L] — BMI was obtained to patients, tear tests and eye measurements were done by primary investigator of the study
  mmol/L
    Native Thiol Mean(Standart Deviation) Unit of measure: mmol/L | 13.96 (38.93) | 2.31 (2.48) | 8.13 (20.70)
    Total Thiol Mean(Standart Deviation) Unit of measure: mmol/L | 34.75 (48.44) | 19.76 (2.93) | 27.25 (25.68)
    Disülfide Mean(Standart Deviation) Unit of measure: mmol/L | 10.76 (6.5) | 8.75 (1.84) | 9.75 (4.17)
BMI [Mean (Standard Deviation); unit: kg/m²] — BMI was obtained to patients
  Mean(Standart Deviation) Unit of measure: kg/m²
  kg/m² | 27.94 (5.28) | 27.76 (5.93) | 27.85 (5.605)
Mean RNFL, Temporal RNFL, CMT [Mean (Standard Deviation); unit: µm] — Eye measurements were done by primary investigator of the study
  µm
    Mean RNFL Mean (standard Deviation) Unit of measure:µm | 101.91 (10.34) | 100.23 (10.87) | 101.07 (10.60)
    RNFL Temporal Mean (standard Deviation) Unit of measure:µm | 80.53 (15.08) | 70.81 (16.43) | 75.67 (15.75)
    CMT Mean (standard Deviation) Unit of measure:µm | 246.59 (19.35) | 252.08 (18.36) | 249.33 (18.85)

OUTCOME MEASURES:

1. Primary Outcome: Glucose Levels of the Groups in Pregnant Women With Impaired Blood Sugar and/or Gestational DM
Description: All patients underwent a 50-g GTT at any time of the day. Women with ≥ 140 mg/dL on the 50-g GTT in the first hour but with a normal 100-g oral GTT level were included in the hyperglycemia group. Women with a 50-g GTT level < 140 mg/dL were categorized as normal and included in the control group
Time Frame: 26 weeks of pregnant
Population: 34 control pregnant women and 26 pregnant women with impaired glucose tolerance were compared with fasting blood glucose and blood glucose at the 1st hour after 50 g sugar loading.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 34 | 26
mg/dl
  50 gr (1hour) Mean(Standart Deviation) Unit of measure: mg/dl | 111.67 (25.54) | 154 (24.29)
  Fasting food sugar Mean(Standart Deviation) Unit of measure: mg/dl | 83.06 (11.33) | 88.15 (14.33)

2. Secondary Outcome: Retinal Nerve Fiber Thickness and Macular Thickness in Pregnant Women With Impaired Blood Sugar and/or Gestational DM
Description: Retinal nerve fiber thickness and macular (µm) are measured by OCT in pregnant women with impaired blood sugar and/or gestational DM RNFL (mean, superior, inferior, nasal, temporal), mean central macular thickness, macula 3mm (mean, superior, inferior, nasal, temporal) and macula 6mm (mean, superior, inferior, nasal, temporal) were measured
Time Frame: 26 weeks pregnant women
Population: Retinal nerve fibre thickness and macular thickness were measured in 26 pregnant women with blood glucose disorders and/or gestational DM and 24 pregnant women in the control group.
Measure: Mean (Standard Error); unit: µm
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 34 | 26
µm
  Mean RNFL Mean(Standart Deviation) Unit of measure:µm | 101.91 (10.34) | 100.23 (10.87)
  Superior RNFL Mean(Standart Deviation) Unit of measure:µm | 123.82 (16.05) | 124.85 (15.78)
  Inferior RNFL Mean(Standart Deviation) Unit of measure:µm | 132.59 (15.92) | 128.23 (20.6)
  Nasal RNFL Mean(Standart Deviation) Unit of measure:µm | 72.12 (10.65) | 72.27 (11.81)
  Temporal RNFL Mean(Standart Deviation) Unit of measure:µm | 80.53 (15.08) | 70.81 (16.43)
  Macula CMT Mean(Standart Deviation) Unit of measure:µm | 246.59 (19.35) | 252.08 (18.36)
  Macula 3mm Superior Mean(Standart Deviation) Unit of measure:µm | 330.5 (14.79) | 333.5 (14.94)
  Macula 3mm Inferior Mean(Standart Deviation) Unit of measure:µm | 326.91 (15.33) | 330.92 (15.33)
  Macula 3mm Nasal Mean(Standart Deviation) Unit of measure:µm | 313.97 (11.98) | 316.88 (17.15)
  Macula 3mm Temporal Mean(Standart Deviation) Unit of measure:µm | 330.88 (13.51) | 330.65 (12.48)
  Macula 6mm Superior Mean(Standart Deviation) Unit of measure:µm | 299.21 (12.36) | 298.19 (12.72)
  Macula 6mm Inferior Mean(Standart Deviation) Unit of measure:µm | 292.32 (22.82) | 285.00 (10.10)
  Macula 6mm Nasal Mean(Standart Deviation) Unit of measure:µm | 280.44 (11.52) | 283.81 (10.26)
  Macula 6mm Temporal Mean(Standart Deviation) Unit of measure:µm | 311.00 (10.88) | 307.92 (12.84)

3. Secondary Outcome: Oxidative Stress Level in Pregnant Women With Impaired Blood Sugar and/or Gestational DM
Description: Native thiol values, total thiol and disulfide values in tears in the pregnant group with blood sugar disorders and/or gestational DM, and control group
Time Frame: 26 weeks of pregnant
Population: Natural thiol values, total thiol and disulphide values in tears of 26 pregnant women with blood glucose disorders and/or gestational DM and 34 control subjects
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 34 | 26
mmol/L
  Native Thiol Mean(Standart Deviation) Unit of measure: mmol/L | 13.96 (38.93) | 2.31 (2.48)
  Total Thiol Mean(Standart Deviation) Unit of measure: mmol/L | 34.75 (48.44) | 19.76 (2.93)
  Disülfide Mean(Standart Deviation) Unit of measure: mmol/L | 10.76 (6.5) | 8.75 (1.84)

4. Secondary Outcome: Retinal Nerve Fiber Temporal Quadrant Thickness in Pregnant Women With Impaired Blood Sugar and/or Gestational DM
Description: Retinal nerve fiber temporal quadrant thickness in the pregnant group with blood sugar disorders and/or gestational DM, and control group
Time Frame: 26 weeks of pregnant
Population: Retinal nerve fibre temporal quadrant thicknesses were measured in tears of 26 pregnant women with blood glucose disorders and/or gestational DM and 34 control subjects.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 34 | 26
µm
  Temporal RNFL Mean(Standart Deviation) Unit of measure:µm | 80.53 (15.08) | 70.81 (16.43)
  Nasal RNFL Mean(Standart Deviation) Unit of measure:µm | 72.12 (10.65) | 72.27 (11.81)
  Superior RNFL Mean(Standart Deviation) Unit of measure:µm | 123.82 (16.05) | 124.85 (15.78)
  Inferior RNFL Mean(Standart Deviation) Unit of measure:µm | 132.59 (15.92) | 128.23 (20.6)

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: Serious Adverse Events is zero. All-Cause Mortality is zero. Other (Not Including Serious) Adverse Events is zero.
Arm/Group | Control Group | Case Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/26
Other Adverse Events (participants affected / at risk) | 0/34 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT05958927/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT05958927/SAP_003.pdf